CLINICAL TRIAL: NCT05983484
Title: Non-Invasive Monitoring of Arrhythmias Electrocardiogram (ECG) Using Textile Sensors (MYANT)
Brief Title: Holter Versus Skiin Garments
Status: Completed | Type: Observational
Sponsor: Myant Medical Corp. (Industry)
Collaborators: Partners in Advanced Cardiac Evaluation (Unknown)
Responsible Party: Sponsor
Other Study IDs: MYANT/PACE - 073-1819-7
Record Dates: First submitted 2023-05-23; First posted 2023-08-09 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Arrhythmia
Keywords: ECG; Wearable; Holter
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Skiin Underwear — All participants enrolled will wear simultaneously the PocketECG (Standard Holter) and the Skiin Underwear Chestband (wearable textile). Each participant will wear both systems for the duration prescribed by their physician (1 to 14 days).
  Other Names: PocketECG

SUMMARY:
The goal of this observational study is to compare the electrocardiogram recording from Holter monitor with textile sensors (in the form of clothing) in patients diagnosed with arrhythmia. The study aims to answer the following questions:

* Can the textile sensors provide continuous monitoring and detect arrhythmias?
* Do patients prefer to wear textile sensors instead of the Holter?

Participants that need Holter monitoring as part of their standard care will be invited to participate in the study. They will simultaneously wear both, the Holter monitor and the textile sensors for the time prescribed by their physician. Participants will also be asked to answer a questionnaire in the initial assessment and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Being addressed to the PACE cardiology clinic to perform an ECG due to a diagnosed or suspected cardiovascular disease.
* Age above 18
* Understand and speak English enough to consent and answer the study questionnaire.
* A medical need for Holter monitoring, and having a personal smartphone (iOS or Android), compatible with the Skiin app (application used to monitor the patient using the wearable device)

Exclusion Criteria:

* Pregnancy
* Implanted defibrillator or pacemaker
* Absence of garment fitting the participant's body
* Open wound or dressing (e.g. band-aid) on a body part that needs to be in contact with the Skiin electrodes
* Severe frailty such that donning or doffing the garment may cause a danger of fall.
* Sensitive skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with cardiovascular disease and/or risks justifying the need for performing an ECG Holter
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Difference in Usable ECG | Throughout the entire data collection period, that is between 1 and 14 days
  The duration of diagnostic ECG from PocketECG minus the duration of diagnostic ECG from Skiin underwear
Difference in Heart Rate | Throughout the entire data collection period, that is between 1 and 14 days
  The heart rate obtained from PocketECG minus the heart rate obtained from Skiin underwear
Difference in RR intervals | Throughout the entire data collection period, that is between 1 and 14 days
  The RR intervals obtained from PocketECG minus the RR intervals obtained from Skiin underwear
Arrhythmic events | Throughout the entire data collection period, that is between 1 and 14 days
  The number and proportion of arrhythmic events obtained by PocketECG and by Skiin underwear

SECONDARY OUTCOMES:
Patient's perception | At the end of the study, 1 to 14 days after initiation.
  A questionnaire developed by Myant containing 10 questions related to the comfort, usability, ease of use and enjoyment will be applied to assess patients' perception of the Skiin underwear and of the PocketECG and to compare both systems, with answers on a 7 point Lickert Scale (from Strongly disagree to Strongly Agree, no numeric scoring).

CONTACTS AND LOCATIONS:
Overall Officials: Yaariv Khaykin, MD, Principal Investigator — Partners in Advanced Cardiac Evaluation
Locations (1):
- Partners in Advanced Cardiac Evaluation (PACE) clinic, Newmarket, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided